CLINICAL TRIAL: NCT03597100
Title: Prospective Study for Symptomatic Relief of Essential Tremor With Cala Therapy
Brief Title: Prospective Study for Symptomatic Relief of ET With Cala Therapy
Acronym: PROSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cala Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET-14
Record Dates: First submitted 2018-06-27; First posted 2018-07-24 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cala TWO (Experimental): Two 40-minute stimulation sessions daily, separated by at least two hours
  Interventions: Device: Cala TWO

INTERVENTIONS:
Device: Cala TWO — Wrist-worn stimulator which applies a tremor-customized stimulation pattern to an individual's nerves

SUMMARY:
Prospective, multi-center, single-arm, non-significant risk study designed to evaluate the Cala TWO device. Subjects will be screened for eligibility and fitted with a Cala TWO device. Subjects will wear the device at home for a period of 3 months, during which they will be asked to stimulate their dominant hand twice a day. The stimulation amplitude will be based on each subject's stimulation threshold. Subjects will have in clinic assessments at enrollment, month 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥22 years of age
* Competent and willing to provide written, informed consent to participate in the study
* A diagnosis of essential tremor as confirmed from clinical history and examination by a movement disorder neurologist
* A tremor severity score of 2 or above in the dominant hand/arm as measured by any one of the TETRAS upper limb items and a minimum subset score of 6 across all upper limb items
* Significant disability due to essential tremor (Bain & Findley score of 3 or above in any one of the upper limb items and a minimum subset score of 8 across all upper limb items)
* Stable dose of tremor medications, if applicable, for 30 days prior to study entry
* Stable dose of antidepressant medications, if applicable, for 90 days prior to study entry
* Willing to comply with study protocol requirements including:

  * remaining on a stable dosage of tremor and antidepressant medications, if applicable, during the duration of the study
  * no significant alcohol or caffeine consumption within 8 hours prior to study visits
  * no usage of the Cala TWO device within 8 hours prior to study visits

Exclusion Criteria:

* Moderate to severe ethanol dependence as defined by the criteria outlined in the DSM-5 (score of 4 or higher)
* Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator, or implanted metal in the wrist to be stimulated
* Previous thalamotomy procedure, including stereotactic thalamotomy, gamma knife radiosurgical thalamotomy, and focused ultrasound for the treatment of tremor
* Suspected or diagnosed epilepsy or other seizure disorder
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
* Peripheral neuropathy affecting the tested upper extremity
* Presence of any other neurodegenerative disease like Parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Anyone suspected to have the diagnosis of idiopathic Parkinson's disease (PD). This includes excluding anyone with the presence of parkinsonian features including bradykinesia rigidity, or postural instability. Subjects who exhibit only mild resting tremor but no other symptoms or signs of PD may be included.
* Botulinum toxin injection for hand tremor within 6 months prior to study enrollment
* Are participating or have participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by the Sponsor
* Significant alcohol or caffeine consumption within 8 hours prior to study enrollment, which may confound the results of the study, where significant caffeine is considered more than 95 mg (equivalent to a cup of coffee), and significant alcohol is considered more than 14 g (equivalent to 5 oz of wine, 12 oz of beer, or 1.5 oz of distilled spirits).
* Subjects unable to communicate with the investigator and staff
* Any health condition that in the investigator's opinion should preclude participation in this study
* Pregnancy or anticipated pregnancy during the course of the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Barrow Neurological Institute (Dignity Health), Phoenix, Arizona
  - USC, Los Angeles, California
  - Parkinson's Institute and Clinical Center, Mountain View, California
  - University of California San Francisco, San Francisco, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - Rocky Mountain Movement Disorders Center, Denver, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Medstar Gerogetown Health Institute, Georgetown, District of Columbia
  - Parkinson's Center, Boca Raton, Florida
  - USF, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Kaiser Mid-Atlantic Group, Largo, Maryland
  - Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, West Bloomfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Advanced Neurology Specialists, Great Falls, Montana
  - Parkinson's Disease and Movement Disorders Center of Long Island, Long Island City, New York
  - Mount Sinai & Beth Isreal, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest, Raleigh, North Carolina
  - River Hills Neuroscience, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University Of Pennsylvania Medicine, Philadelphia, Pennsylvania
  - Jefferson University, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Texas Movement Disorder Specialist, Georgetown, Texas
  - Houston Methodist, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Swedish, Bellevue, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cala TWO
Started | 263
Completed | 205
Not Completed | 58

BASELINE CHARACTERISTICS:
Arm/Group | Cala TWO
Number analyzed (Participants) | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 253
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 237
  More than one race | 3
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 263

OUTCOME MEASURES:

1. Primary Outcome: TRG (Tremor Research Group) Essential Tremor Rating Assessment Scale (TETRAS) Subset Score
Description: Tremor Research Group (TRG) Essential Tremor Rating Assessment Scale (TETRAS) subset score: TETRAS subset score relevant to the stimulated upper limb. The subset score is the sum of 6 rated tasks. Each task is rated 0 to 4, where a higher score indicates more severe tremor. Minimum subset score = 0; Maximum subset score = 24.
Time Frame: Baseline to 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cala TWO
Number analyzed (Participants) | 205
score on a scale
  Baseline | 12.6 (2.7)
  Final Visit | 9.8 (3.5)
  Change | -2.8 (2.8)

2. Primary Outcome: Bain & Findley Activities of Daily Living (ADL) Scale Subset Score
Description: Bain & Findley ADL subset score relevant to the stimulated upper limb. The subset score is the sum of 8 rated tasks. Each task is rated 1 to 4, where a higher score indicates more severe tremor. Minimum subset score = 8; Maximum subset score = 32.
Time Frame: Baseline to 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cala TWO
Number analyzed (Participants) | 205
score on a scale
  Baseline | 18.4 (3.8)
  Final Visit | 13.4 (4.4)
  Change | -4.98 (4.3)

3. Secondary Outcome: Kinematic Measurements, as Collected With the Device During Postural Holds, Change From Pre-stimulation to Post-stimulation Across Sessions
Description: Subjects will be prompted to perform a postural hold task before and after each stimulation session. During this task, the device will record kinematic data using on-board motion sensors to objectively assess if there are any changes in tremor level. The change in each patient's pre- and post-stimulation tremor power was defined as the median change over all valid stimulation sessions. Sample mean and standard deviations were computed using the median change value from all patients.
Time Frame: Average change in tremor power over 3-month study period
Measure: Mean (Standard Deviation); unit: (m/s^2)^2
Arm/Group | Cala TWO
Number analyzed (Participants) | 193
(m/s^2)^2 | -0.8 (3.7)

ADVERSE EVENTS:
Time Frame: Up to 3 months since baseline testing
Arm/Group | Cala TWO
All-Cause Mortality (participants affected / at risk) | 1/263
Serious Adverse Events (participants affected / at risk) | 5/263
Other Adverse Events (participants affected / at risk) | 47/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cala TWO (N=263)
Initial or prolonged hospitalization (General disorders) | 5 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cala TWO (N=263)
Significant and persistent skin irritation (Skin and subcutaneous tissue disorders) | 14 (15)
Sore/Lesion (Skin and subcutaneous tissue disorders) | 10 (11)
Significant discomfort (Skin and subcutaneous tissue disorders) | 6 (7)
Electrical burns (Skin and subcutaneous tissue disorders) | 6 (6)
Minor Skin Irritation (Skin and subcutaneous tissue disorders) | 6 (6)
Electric shock sensation while using device (Skin and subcutaneous tissue disorders) | 3 (3)
Worsening of tremor (Nervous system disorders) | 2 (2)
Other isolated events (Skin and subcutaneous tissue disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03597100/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03597100/SAP_002.pdf